CLINICAL TRIAL: NCT01721265
Title: 3-Year, Observational Study to Evaluate the Durability of Sustained Viral Response and the Kinetics of Antiviral-Resistant HCV in Subjects Who Participated in Studies of Idenix Anti-HCV, Direct Acting Antivirals
Brief Title: 3-Year Observational Virology Follow-up Study in Subjects Who Participated in Studies of Idenix Anti-HCV, Direct Acting Antivirals
Status: Terminated | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 1894-009; IDX-03YF
Record Dates: First submitted 2012-10-31; First posted 2012-11-05 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Hepatitis C
Keywords: HCV; Hepatitis C; IDX184; IDX719
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
All subjects in this study have previously been in an Idenix HCV study and received study drug for 3 consecutive days. Subjects who had received placebo in a previous Idenix study will not be enrolled in this study.

In this study, researchers will try to find answers to these questions:

* How much (if any) hepatitis C virus is in your blood after stopping your Idenix study drug?
* Is your hepatitis C virus possibly resistant to treatment with the Idenix study drug or similar drugs?

DETAILED DESCRIPTION:
The data obtained from this study will be used to further understand the long-term efficacy of Idenix DAAs used to treat HCV infection and to further understand HCV resistance to Idenix DAAs.

ELIGIBILITY:
Inclusion Criteria:

* Read and signed the written informed consent form (ICF) after the nature of the study has been fully explained
* Have participated in an Idenix-sponsored study of an Idenix DAA
* Received at least 3 consecutive days of DAA treatment in an Idenix-sponsored study
* Agreed to comply with the visit schedule and laboratory tests

Exclusion Criteria:

* Treatment with placebo only, in an Idenix sponsored study
* Antiviral treatment for HCV after participation in an Idenix sponsored study of an Idenix DAA

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will include subjects who participated in studies of Idenix anti-HCV DAAs.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2012-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Durability of Sustained viral response [SVR] | every 3 months
  To evaluate the durability of sustained virological response (SVR). Plasma HCV RNA levels will be monitored over time.

SECONDARY OUTCOMES:
Kinetics of resistant variants | every 3 months
  To describe the kinetics of resistant variants to Idenix direct acting antivirals (DAAs) by HCV RNA sequencing. The presence of each identified resistant variant in the viral population will be descriptively evaluated until the viral population consists entirely of wild-type virus or over a period of 3 years, whichever comes first.